CLINICAL TRIAL: NCT02419976
Title: Electronic Nose Identification of Fasting and Non-fasting Breath Profiles
Acronym: Fast Breath
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a loss of funding and all activities in the Netherlands being terminated as of June 20th 2024. IP & assets belong to eNose Holding BV.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Cadman Leggett, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 14-009226
Record Dates: First submitted 2015-04-07; First posted 2015-04-17 (Estimated); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Breath Analysis (Experimental): Individuals consenting to participation of this study will be asked to provide a breath analysis using the Aeonose. Following their scheduled standard of care endoscopic procedure the patient will repeat the breath analysis.
  Interventions: Other: a breath analysis using the Aeonose; Device: Aeonose

INTERVENTIONS:
Other: a breath analysis using the Aeonose — using the Aeonose per standard acquisition protocol which spans 15 minutes of which the individuals breaths normally through a sterile disposable mouthpiece with sterile disposable air filters for 5 minutes during signal acquisition while wearing a nose plug. This will be completed in the office setting prior to their endoscopic procedure.
  Following their scheduled standard of care endoscopic procedure the patient will be allowed to consume a standardized refreshment (such as juice or soda) prior to discharge from the post procedure area. These refreshments are already provided as standard care. The participant will return to the office setting and repeat the same breath analysis acquisition process that was done prior to the procedure.
  Other Names: Enose
Device: Aeonose

SUMMARY:
The investigators will study a noninvasive no risk process by which the investigators can quickly screen and assess for fasting and non-fasting states in individuals scheduled for routine endoscopy.

DETAILED DESCRIPTION:
The investigators will study a noninvasive no risk process by which we can quickly screen and assess for fasting and non-fasting states in individuals scheduled for routine endoscopy. In non-fasting individuals, the risk of a sedation related complication such as aspiration increases and often the procedure must be aborted and repeated on another day following more prolonged fasting and medication administration. This adds to increased cost and delay to patient care.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Adult (18+) patient undergoing scheduled elective outpatient upper endoscopy
  2. Willing and able to consent to research protocol
  3. Fasting as required per routine instruction for upper endoscopy
  4. Able to breath for approximately 10 minutes pre and post procedure into the Aeonose device with a nose-plug on
  5. Able to consume standard refreshments post procedure during recovery per routine endoscopic area policy

     Exclusion Criteria:

  <!-- -->

  1. Non-fasting per protocol, or known to have had food or drink outside of routine protocol
  2. < 18 years of age
  3. Unable or unwilling to consent to research protocol
  4. Inability to tolerate Aeonose breathing (such as those with claustrophobia, anxiety, nasal trauma, etc.)
  5. Unable to consume refreshment post procedurally
  6. Unable to repeat Aeonose measurement post-procedurally due to tolerance or medical indication (such as instructed to remain fasting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2015-02; Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cadman Leggett, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol required classifying subjects as fasting or non-fasting, but only 185 fasting and 33 non-fasting subjects can be reported. As the data field in the study database designated to record fasting status was not implemented consistently throughout the study, fasting information was as a result not collected for the majority of enrolled subjects. The study team cannot retrospectively determine or report fasting status for the remaining subjects.
Groups:
- Fasting Breath Analysis: Individuals consenting to participation of this study will be asked to provide a breath analysis using the Aeonose. Following their scheduled standard of care endoscopic procedure the patient will repeat the breath analysis
  a breath analysis using the Aeonose: using the Aeonose per standard acquisition protocol which spans 15 minutes of which the individuals breaths normally through a sterile disposable mouthpiece with sterile disposable air filters for 5 minutes during signal acquisition while wearing a nose plug. This will be completed in the office setting prior to their endoscopic procedure.
  Following their scheduled standard of care endoscopic procedure the patient will be allowed to consume a standardized refreshment (such as juice or soda) prior to discharge from the post procedure area. These refreshments are already provided as standard care. The participant will return to the office setting and repeat the same breath analysis acquisition process that was done prior to the procedure.
  Aeonose
Period: Overall Study
Arm/Group | Fasting Breath Analysis
Started | 879
Fasting | 185
Non-Fasting | 33
Completed | 879
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fasting Breath Analysis: Individuals consenting to participation of this study will be asked to provide a breath analysis using the Aeonose. Following their scheduled standard of care endoscopic procedure the patient will repeat the breath analysis
  a breath analysis using the Aeonose: using the Aeonose per standard acquisition protocol which spans 15 minutes of which the individuals breaths normally through a sterile disposable mouthpiece with sterile disposable air filters for 10 minutes during signal acquisition while wearing a nose plug. This will be completed in the office setting prior to their endoscopic procedure.
  Following their scheduled standard of care endoscopic procedure the patient will be allowed to consume a standardized refreshment (such as juice or soda) prior to discharge from the post procedure area. These refreshments are already provided as standard care. The participant will return to the office setting and repeat the same breath analysis acquisition process that was done prior to the procedure.
  Aeonose
Arm/Group | Fasting Breath Analysis
Number analyzed (Participants) | 879
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 456
  >=65 years | 423
Age, Continuous [Mean (Full Range); unit: years] | 44 [18 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 331
  Male | 548
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 780
  Unknown or Not Reported | 89
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 786
  More than one race | 0
  Unknown or Not Reported | 77
Region of Enrollment [Number; unit: participants]
  United States | 879

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of the Aeonose in Distinguishing a Fasting Versus Non-fasting Breath Profile
Description: Exhaled Volatile Organic Compounds (VOCs) were collected by subject's breathing into a non-invasive breath analyzer (Aeonose) for 5 minutes by which through pattern recognition electronic changes can be identified in exhaled volatile organic compounds interfacing with an electronic sensor that creates an electronic signature, or smell-print that distinguishes the fasting and non-fasting states. The effectiveness of the Aeonose in distinguishing subjects in a fasting versus non-fasting state is represented by the device's sensitivity and specificity (ability to positively identify subjects who are in a fasting state versus non-fasting state).
Time Frame: breath analysis obtained (approximately 10 minutes procedure)
Population: Due to loss of funding and the closure of the device provider, the study team was unable to obtain or access the device-generated data on 661 subjects. As a result, this data was never uploaded to the study database and cannot be retrieved.
Measure: Count of Participants; unit: Participants
Groups:
- Breath Analysis: Individuals consenting to participation of this study will be asked to provide a breath analysis using the Aeonose. Following their scheduled standard of care endoscopic procedure the patient will repeat the breath analysis a breath analysis using the Aeonose: using the Aeonose per standard acquisition protocol which spans 15 minutes of which the individuals breaths normally through a sterile disposable mouthpiece with sterile disposable air filters for 5 minutes during signal acquisition while wearing a nose plug. This will be completed in the office setting prior to their endoscopic procedure.
  Following their scheduled standard of care endoscopic procedure the patient will be allowed to consume a standardized refreshment (such as juice or soda) prior to discharge from the post procedure area. These refreshments are already provided as standard care. The participant will return to the office setting and repeat the same breath analysis acquisition process that was done prior to the procedure.
  Aeonose
Arm/Group | Breath Analysis
Number analyzed (Participants) | 218
Participants
  Sensitivity | 194
  Specificity | 185
  Accuracy | 194
  Positive Predictive Value | 212
  Negative Predictive Value | 126

ADVERSE EVENTS:
Time Frame: N/A because participants were not monitored/assessed for adverse events during the study
Description: There were no tracked adverse events or risks because it was a minimum risk breath test prior to an EGD procedure. The participants were not at risk of any Serious adverse Events or All-Cause mortality.
Groups:
- Non Fasting Breath Analysis: Individuals consenting to participation of this study will be asked to provide a breath analysis using the Aeonose. Following their scheduled standard of care endoscopic procedure the patient will repeat the breath analysis
  a breath analysis using the Aeonose: using the Aeonose per standard acquisition protocol which spans 15 minutes of which the individuals breaths normally through a sterile disposable mouthpiece with sterile disposable air filters for 10 minutes during signal acquisition while wearing a nose plug. This will be completed in the office setting prior to their endoscopic procedure.
  Following their scheduled standard of care endoscopic procedure the patient will be allowed to consume a standardized refreshment (such as juice or soda) prior to discharge from the post procedure area. These refreshments are already provided as standard care. The participant will return to the office setting and repeat the same breath analysis acquisition process that was done prior to the procedure.
  Aeonose
Arm/Group | Non Fasting Breath Analysis
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated early due to a loss of funding and all activities in the Netherlands being terminated as of June 20th 2024.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT02419976/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02419976/ICF_001.pdf